CLINICAL TRIAL: NCT02408354
Title: "Etude Pilote, Comparative, Monocentrique, randomisée, en Cross Over, en Double Aveugle, Contre Placebo, Testant l'efficacité de l'Huile triheptanoïne Dans Les Hémiplégies Alternantes de l'Enfant" HEMIHEP
Brief Title: Pilot Study, Comparative, Single-center, Randomized, Crossover, Double-blind, Against Placebo, Testing the Effectiveness of Triheptanoin Oil in Alternating Hemiplegia of Childhood
Acronym: HEMIHEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C14-53
Record Dates: First submitted 2015-03-24; First posted 2015-04-03 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Alternating Hemiplegia of Childhood
MeSH Terms: conditions — Alternating hemiplegia of childhood | interventions — triheptanoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triheptanoin (Active Comparator): Triheptanoin/ Placebo Randomized to receive active Triheptanoin first for 12 weeks. At cross-over, participants will receive placebo for 12 weeks.
  Each drug will be dispensed successively. A one-month wash out period is planned for 4 weeks between triheptanoine and placebo phases.
  Interventions: Drug: Triheptanoin
- Placebo (Placebo Comparator): Placebo / Triheptanoin Randomized to receive active Placebo first for 12 weeks. At cross-over, participants will receive Triheptanoin for 12 weeks.
  Each drug will be dispensed successively. A one-month wash out period is planned for 4 weeks between placebo and triheptanoin phases.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Triheptanoin — Triheptanoin is a triglyceride composed of three heptanoate (C7 fatty acid) esters. Triheptanoin is manufactured by chemical synthesis from glycerol and heptanoic acid. Triheptanoin is a liquid, intended for oral (PO) administration.
  Participants will be given approximately 1g/kg of Triheptanoin divided at least in three doses (at 8 am, 12 noon, and 8 pm). A one-day titration period will be used, using 0.5 g/kg increments before arriving at the full dose.
  Other Names: UX007; glycerol triheptanoate
  Arms: Triheptanoin
Drug: Placebo — Placebo is a oily liquid, intended for oral (PO) administration. Participants will be given approximately 1g/kg of Placebo divided at least in three doses (at 8 am, 12 noon, and 8 pm). A one-day titration period will be used, using 0.5 g/kg increments before arriving at the full dose.
  Arms: Placebo

SUMMARY:
The purpose of this project is to study the efficacy of triheptanoin oil in patients with Alternating Hemiplegia of Childhood (AHC) due to ATP1A3 gene mutation.

DETAILED DESCRIPTION:
The clinical spectrum of Alternating Hemiplegia of Childhood (AHC) is wide and characterized by the association of permanent and paroxysmal (palsy, dystonia, ocular, epileptic, dysautonomic events) neurological events, with onset in childhood. Most of AHC patients carry mutations in the ATP1A3 gene. This gene encodes the Na+/K+ ATPase witch is a transmembrane ion pump generating chemical and electrical gradient of sodium and potassium across the plasma membrane. Those paroxystic events in AHC patients with mutations in the ATP1A3 gene could be associated with a glucidic/energetic metabolism or intracerebral excitability disorder.

Triheptanoin is a triglyceride, whose derivatives pass the blood - brain barrier and enhance the Krebs cycle functions. Triheptanoin could therefore allow energy supply to the brain, which is essential for the functioning of the Na+/ K+ ATPase that consumes a significant amount of energy in the brain.

The investigators goal is to do a pilot study to test the effectiveness on paroxystic manifestations and the safety of triheptanoin in a small group of patients with Alternating Hemiplegia of Childhood secondary to ATP1A3 mutations.

ELIGIBILITY:
Inclusion Criteria:

* AHC with mutation in ATP1A3 gene
* Age ≥ 15 years and 3 months
* ≥ 6 neurological paroxystic events during the last 3 months prior to the beginning of the study
* No specific diet
* Covered by french social security
* Patients who freely agree to participate in this study and understand the nature, risks and benefits of this study and give their written informed consent. (In addition to the requirement for the consent of parents or the legal representative, adolescents can provide additional informed consent to participate in clinical trials)

Exclusion Criteria:

* Age < 15 years and 3 months
* Evidence of psychiatric disorder
* Comorbid medical condition that would render them unsuitable for the study, e.g. HIV, diabetes
* Pregnant or parturient or lactating women
* Absence of double effective contraception at the women old enough to procreate
* Unwillingness to be informed in case of abnormal MRI
* Absence of signed informed consent
* No covered by french social security
* Persons deprived of their liberty by judicial or administrative decision
* Person subject to an exclusion period for another research
* Subjects with exclusion criteria required by french law

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Number of neurologic paroxystic events report in patient diary | 7 months
  visit 1 at day 0, visit 2 at week 12, visit 3 at week 16, visit 4 at week 28

SECONDARY OUTCOMES:
Composite score allying the number of neurological paroxystic events, their duration and severity. | 7 months
  visit 1 at day 0, visit 2 at week 12, visit 3 at week 16, visit 4 at week 28
Clinical Global Impression Scales - Improvement | 7 months
  visit 2 at week 12, visit 4 at week 28
The Short Form (36) Health Survey | 7 months
  visit 1 at day 0, visit 2 at week 12, visit 3 at week 16, visit 4 at week 28
Brain 31phosphorus magnetic resonance spectroscopy | 7 months
  Ratio of Inorganic Phosphate (Pi) over Phosphocreatine during visual stimulation visit 2 at week 12, visit 4 at week 28
Clinical Safety as measured by questionnaire | 7 months
  visit 2 at week 12, visit 4 at week 28
Biological Safety as measured by acylcarnitine profile, organic acid dosage | 7 months
  visit 2 at week 12, visit 4 at week 28

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Flamand-Roze, MD, PhD, Principal Investigator — INSERM UMRS 975, 47 bd de l'hôpital - 75651 Paris Cedex 13
Locations (1):
- Groupe hospitalier Pitié Salpêtrière, Paris, France

REFERENCES:
- [Result] Hainque E, Caillet S, Leroy S, Flamand-Roze C, Adanyeguh I, Charbonnier-Beaupel F, Retail M, Le Toullec B, Atencio M, Rivaud-Pechoux S, Brochard V, Habarou F, Ottolenghi C, Cormier F, Meneret A, Ruiz M, Doulazmi M, Roubergue A, Corvol JC, Vidailhet M, Mochel F, Roze E. A randomized, controlled, double-blind, crossover trial of triheptanoin in alternating hemiplegia of childhood. Orphanet J Rare Dis. 2017 Oct 2;12(1):160. doi: 10.1186/s13023-017-0713-2. PMID 28969699